CLINICAL TRIAL: NCT00004183
Title: Capecitabine (Xeloda) in Malignant Mesothelioma: A Phase II Study
Brief Title: Capecitabine in Treating Patients With Malignant Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-39807; U10CA031946 (NIH); CLB-39807; CDR0000067422 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2000-01-21; First posted 2004-02-25 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Malignant Mesothelioma
Keywords: localized malignant mesothelioma; advanced malignant mesothelioma; recurrent malignant mesothelioma; epithelial mesothelioma; sarcomatous mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant; Solitary Fibrous Tumor, Pleural | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- capecitabine (Experimental): Patients receive oral capecitabine twice daily on days 1-14. Treatment repeats every 3 weeks for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 2 months for 1 year, every 3 months for 2 years and then annually thereafter.
  Interventions: Drug: capecitabine

INTERVENTIONS:
Drug: capecitabine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of capecitabine in treating patients who have malignant mesothelioma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate, overall survival, and failure free survival of patients with malignant mesothelioma treated with capecitabine. II. Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients receive oral capecitabine twice daily on days 1-14. Treatment repeats every 3 weeks for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 2 months for 1 year, every 3 months for 2 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study within 7-9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven malignant mesothelioma not amenable to potentially curative radiotherapy or surgery Epithelial, sarcomatoid, or mixed subtype Any site of origin allowed including, but not limited to, the following: Pleura Peritoneum Pericardium Tunica vaginalis Measurable disease At least one lesion accurately measured in at least one dimension Lesion at least 20 mm at largest diameter with conventional techniques or at least 10 mm with spiral CT scan The following are not considered measurable disease: Bone lesions Leptomeningeal disease Ascites Pleural/pericardial effusion Abdominal masses not confirmed and followed by imaging techniques Cystic lesions Tumor lesions located in a previously irradiated area

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0 or 1 Life expectancy: Not specified Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT no greater than 2.5 times ULN Renal: Creatinine no greater than 1.5 times ULN Other: Not pregnant or nursing Fertile patients must use effective contraception No active second malignancy except nonmelanomatous skin cancer Not considered an active second malignancy if: Therapy has been completed Less than 30% risk of relapse according to the physician No malabsorption syndrome

PRIOR CONCURRENT THERAPY: Biologic therapy: Concurrent epoetin alfa allowed Chemotherapy: No prior systemic cytotoxic chemotherapy for malignant mesothelioma Prior intrapleural cytotoxic or sclerosing agents (including bleomycin) allowed No other concurrent chemotherapy Endocrine therapy: No concurrent hormonal therapy except the following: Steroids administered for adrenal failure Hormonal therapy administered for nonmalignant conditions (e.g., insulin for diabetes) Intermittent use of dexamethasone as an antiemetic Radiotherapy: At least 4 weeks since prior radiotherapy Prior irradiation of symptomatic lesion allowed if there is other measurable disease outside the radiation port No concurrent radiotherapy Surgery: At least 2 weeks since prior major surgery Other: No concurrent leucovorin calcium or folinic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2000-11; Primary Completion 2003-12 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Otterson, MD, Study Chair — Ohio State Comprehensive Cancer Center
Locations (50):
- United States (50):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - University of California San Diego Cancer Center, La Jolla, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Illinois at Chicago Health Sciences Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Veterans Affairs Medical Center - Togus, Togus, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - CCOP - Southwestern Vermont Regional Cancer Center, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Result] Otterson GA, Herndon JE 2nd, Watson D, Green MR, Kindler HL; Cancer and Leukemia Group B. Capecitabine in malignant mesothelioma: a phase II trial by the Cancer and Leukemia Group B (39807). Lung Cancer. 2004 May;44(2):251-9. doi: 10.1016/j.lungcan.2003.10.011. PMID 15084390
- [Result] Otterson GA, Herndon J, Watson D, et al.: Capecitabine in malignant mesothelioma: a phase II trial by the Cancer and Leukemia Group B (CALGB 39807). [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-2778, 691, 2003.